CLINICAL TRIAL: NCT05830513
Title: OPU-LUX: Virtual Reality for Pain and Anxiety Management During Oocyte Pick-up - a Randomized Controlled Trial
Brief Title: OPU-LUX: Virtual Reality for Pain and Anxiety Management During Oocyte Pick-up
Acronym: OPU-LUX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPU-LUX
Record Dates: First submitted 2023-03-14; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-03

CONDITIONS: Pain, Postoperative; IVF
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Women will be randomly allocated to undergo OPU either with the use of Virtual reality(group A)
  Interventions: Device: Virtual Reality
- Group B (No Intervention): Women will be randomly assigned to an OPU in the control group with standard treatment, withouth analgesia (Group B).

INTERVENTIONS:
Device: Virtual Reality — Women will be randomly allocated to undergo OPU either with the use of virutal reality (group A) or the control group with standard treatment, without analgesia(group B). The participants of group A will wear the Oculus Quest 2 and will be surrounded by a virtual world. They will see objects flying towards themselves. They will be able to interact with the virtual world by hand controllers and can try to catch the objects.
  Arms: Group A

SUMMARY:
In vitro fertilization (IVF) cycles are increasingly performed worldwide. Transvaginal oocyte pick-up (OPU) is a painful part of IVF. OPU in polyfollicular IVF is usually performed under sedation and pain relief. In natural cycle IVF or IVF with minimal stimulation OPU is possible without anesthesia. Mostly of the women reported experiencing mild to moderate pain when undergoing OPU without anesthesia. Nevertheless, there is a need for alternative pain treatment options during OPU to reduce the burden of IVF for patients. Virtual reality (VR) may have a role in acutely painful procedures as a non-pharmacological alternative. VR refers to the interactions between an individual and a computer-generated environment stimulating multiple sensory modalities. The immersive, entertaining effects of VR could be useful for redirecting the patient's attention away from painful treatment experiences and reducing anxiety, discomfort, or unpleasantness. Use of VR interventions has been studies in a wider range of medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 43 years
* IVF with follicular aspiration of one to tree follicles
* Written informed consent signed by the participant must be obtained prior to OPU

Exclusion Criteria:

* OPU with more than tree follicular aspiration
* Individuals' anatomy complicating the intervention (e. g. endometriosis stage III/IV)
* Application of analgesics within eight hours before OPU
* hearing impairments
* migraines
* seizure disorder
* vestibular abnormalities
* history of motion sickness

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
VAS | post OPU (line from 0: no pain to 10:worst pain) immediately post OPU
  visual analogue scale pain scoring

SECONDARY OUTCOMES:
VAS for anxiety | Pre-post OPU (line from 0: no to 10:worst anxiety) pre- und immediately post OPU
  VAS for anxiety
state-trait anxiety inventory form (STAI) | Pre-OPU
  state-trait anxiety inventory form (STAI)
vital parameters: pulse rate | Intraoperative
  vital parameters : pulse rate
vital parameters: blood pressure | Intraoperative
  vital parameters: blood pressure (systolic and diastolic pressures)
vital parameters : oxygen saturation | Intraoperative
  vital parameters : oxygen saturation

CONTACTS AND LOCATIONS:
Locations (1):
- PD. Dr. med. Kohl Schwartz, Alexandra, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided